CLINICAL TRIAL: NCT06550765
Title: Safety and Efficacy of Degradable Magnesium Metal Clips in Surgical Margins of Radical Surgery for Malignant Bone and Soft Tissue Tumors: A Single-Center, Randomized Controlled Study
Brief Title: Safety and Efficacy of Degradable Magnesium Metal Clips in Surgical Margins of Radical Surgery for Malignant Bone and Soft Tissue Tumors
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PureMgBoneCuttingEdge
Record Dates: First submitted 2024-07-21; First posted 2024-08-13 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-07

CONDITIONS: Sarcoma, Soft Tissue; Sarcoma, Spindle Cell
Keywords: Soft Tissue sarcoma; biodegradable magnesium metal
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Intervention Model Description: Experimental Group: The tumor lesion area is exposed using conventional methods, and the tumor segment is resected according to the principles of tumor-free operation. Magnesium metal closure clips are used to clamp the tumor blood vessels, osteoperiosteal bleeding points, and other bleeding sites. The lesion area is thoroughly rinsed to ensure no active bleeding, and routine necessary reconstruction is performed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): The tumor lesion area is exposed using conventional surgery methods, and the tumor segment is resected according to the principles of tumor-free operation. Electrocautery and suture ligation are used to handle the tumor bleeding sites. The lesion area is thoroughly rinsed to ensure no active bleeding, and routine necessary reconstruction is performed.
- Magnesium metal closure clips (Experimental): The tumor lesion area is exposed using conventional methods, and the tumor segment is resected according to the principles of tumor-free operation. Magnesium metal closure clips are used to clamp the tumor blood vessels, osteoperiosteal bleeding points, and other bleeding sites. The lesion area is thoroughly rinsed to ensure no active bleeding, and routine necessary reconstruction is performed.
  Interventions: Device: Biodegradable Magnesium Metal Clips

INTERVENTIONS:
Device: Biodegradable Magnesium Metal Clips — The tumor lesion area is exposed using conventional methods, and the tumor segment is resected according to the principles of tumor-free operation. Magnesium metal closure clips are used to clamp the tumor blood vessels, osteoperiosteal bleeding points, and other bleeding sites. The lesion area is thoroughly rinsed to ensure no active bleeding, and routine necessary reconstruction is performed.
  Arms: Magnesium metal closure clips

SUMMARY:
To verify and evaluate the safety and efficacy of biodegradable magnesium metal clips in the surgical margins of radical surgery for bone and soft tissue malignant tumors.

DETAILED DESCRIPTION:
The purpose of this study is to verify and evaluate the safety and effectiveness of biodegradable magnesium metal clips in the surgical margins of radical surgery for bone and soft tissue malignant tumors. The study will be divided into two groups:

Experimental Group: The tumor lesion area is exposed using conventional methods, and the tumor segment is resected according to the principles of tumor-free operation. Magnesium metal closure clips are used to clamp the tumor blood vessels, osteoperiosteal bleeding points, and other bleeding sites. The lesion area is thoroughly rinsed to ensure no active bleeding, and routine necessary reconstruction is performed.

Control Group: The tumor lesion area is exposed using conventional methods, and the tumor segment is resected according to the principles of tumor-free operation. Electrocautery and suture ligation are used to handle the tumor bleeding sites. The lesion area is thoroughly rinsed to ensure no active bleeding, and routine necessary reconstruction is performed.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be of either gender, aged between 18 and 65 years;
2. Diagnosis must be confirmed pathologically as osteosarcoma, synovial sarcoma, liposarcoma, or other bone and soft tissue sarcomas;
3. Must have undergone standard chemotherapy and require en bloc resection;
4. Participants must voluntarily enroll and sign an informed consent form; willing to closely cooperate with the physician to comply with all study requirements, including participation in all follow-up and assessments.

Exclusion Criteria:

1. Severe dysfunction of the heart, liver, kidney, lung, or brain.
2. Pregnant women or women who are breastfeeding.
3. History of autoimmune disease, HIV infection, history of immunosuppressive disorder, or currently taking immunosuppressive drugs.
4. History of syphilis (Treponema pallidum), active infection with hepatitis B or C, and positive for verified antigens.
5. Participation in any other clinical study currently or within 3 months prior to the screening visit.
6. Patients have any other conditions that the researcher deems unsuitable for the study. Age is between 18 to 75 years old.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2024-08-25 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
1-year tumor recurrence rate | 1 year
  Calculate the recurrence rate of the tumor one year after surgery.
Total drainage volume | on the first, second, third, and fourth postoperative days.
  Placement of a drainage tube in the surgical area, with postoperative drainage volumes recorded on the first, second, third, and fourth days.

SECONDARY OUTCOMES:
Blood magnesium ions levels | at one month and six months after the operation
  Measure the magnesium ions levels in the blood before surgery, one month after surgery, and six months after surgery.
  Magnesium ions in the blood are measured in mmol/L. The normal range of serum magnesium is 0.75 to 1.25 mmol/L. Hypermagnesemia is defined as serum magnesium levels greater than 1.25 mmol/L, and hypomagnesemia is defined as serum magnesium levels less than 0.75 mmol/L. Assess the impact of the degradation of the biodegradable enzyme-metal clip on the magnesium ions in the blood, and thereby evaluate its safety for the human body.
Serum alanine aminotransferase (ALT) | at one month and six months after the operation
  Venous blood is collected and sent to Guangdong Provincial People's Hospital Department of Laboratory Medicine for analysis one month and six months after surgery.
  The normal range of serum alanine aminotransferase (ALT) is 7 to 40 U/L. When ALT is beyond the normal range, we consider that the biodegradable magnesium metal clip has caused liver damage during its degradation process, thus evaluating the safety of the metal clip.
Serum creatinine | at one month and six months after the operation
  For normal renal function, the serum creatinine levels are 0.6 - 1.2 mg/dL (53 - 106 µmol/L) for adult males and 0.5 - 1.1 mg/dL (44 - 97 µmol/L) for adult females. Mild renal impairment is indicated by serum creatinine levels of 1.3 - 1.9 mg/dL (115 - 168 µmol/L) in males and 1.2 - 1.8 mg/dL (106 - 159 µmol/L) in females. Moderate renal impairment is reflected by levels of 2.0 - 4.0 mg/dL (177 - 354 µmol/L) in males and 1.9 - 4.0 mg/dL (168 - 354 µmol/L) in females. Severe renal impairment is indicated by serum creatinine levels of 4.1 - 8.0 mg/dL (362 - 707 µmol/L) for both genders. End-stage renal disease (ESRD) is classified by serum creatinine levels greater than 8.0 mg/dL (>707 µmol/L) for both genders. These classifications may vary based on specific clinical standards or guidelines and should be considered in conjunction with other clinical indicators and professional medical judgment.
Estimated glomerular filtration rate (eGFR） | at one month and six months after the operation
  The estimated glomerular filtration rate (eGFR) is a key indicator of kidney function, used to classify chronic kidney disease (CKD) into different stages:
  Stage 1: eGFR ≥ 90 mL/min/1.73 m², indicating normal kidney function. Stage 2: eGFR 60-89 mL/min/1.73 m², representing mildly decreased kidney function.
  Stage 3: Divided into two sub-stages:
  Stage 3a: eGFR 45-59 mL/min/1.73 m², indicating moderate kidney impairment. Stage 3b: eGFR 30-44 mL/min/1.73 m², reflecting more significant kidney dysfunction.
  Stage 4: eGFR 15-29 mL/min/1.73 m², showing severe kidney impairment. Stage 5: eGFR < 15 mL/min/1.73 m² or requiring dialysis, indicating kidney failure.
  These eGFR values help in evaluating kidney function and determining the appropriate treatment approach, with specific adjustments based on clinical guidelines and individual patient factors.

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong provincial people's hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
Researchers can request access from the corresponding author upon reasonable inquiry.